CLINICAL TRIAL: NCT03205631
Title: Comparison of the Natural Frequencies Technology Sleep Patches to Sham Patches During Sleep in the Home Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IC-IT Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NFT-001
Record Dates: First submitted 2017-06-29; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Natural Frequency Patch (Sham Comparator)
  Interventions: Other: Natural Frequency Patch
- Active Natural Frequency Patch (Active Comparator)
  Interventions: Other: Natural Frequency Patch

INTERVENTIONS:
Other: Natural Frequency Patch — Participants will receive in randomized order the differing patches to wear during three nights separated by a washout period of 3-4 nights

SUMMARY:
Prospective, randomized crossover study to compare the NFT sleep patches to sham device to assess sleep via home sleep testing device in the home environment

ELIGIBILITY:
Inclusion Criteria:

* capacity to provide informed consent
* BMI <30
* between 30 and 65 years old
* in overall good health as determined by history and physical assessment subjects pre-screened to ensure they are drug free
* work a typical day job/work week.
* not traveled > 3 time zones in the last month
* typical bedtime between 9-12 PM
* estimated on average 6 hours per night
* negative urine drug screen
* have self-reported unrefreshing sleep for the past month
* agree to limit alcohol use to no more than two drinks a night during the testing period and four hours prior to bedtime
* agree to limit caffeine consumption to four hours prior to bedtime
* ≤ 2 on the depression scale
* ≤ 3 on the anxiety scale

Exclusion Criteria:

* pregnant or nursing a child
* self-induced short sleep habits (<6 hours per night)
* unstable medical conditions as determined by the clinician
* current sleep disorder (sleep apnea AHI/REI<5, restless legs, periodic limb movements, narcolepsy)
* self-reported sleep latency of >30 minutes or early (3-4 AM) awakenings on a regular basis
* contact dermatitis to adhesives
* excluded Medications: over the counter sleep aids, prescribed sleep aids, central nervous system stimulants, antidepressants, sedating antihistamines, over the counter decongestants and opioids

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-06-26 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | three nights
  Assess sleep via home EEG recording

CONTACTS AND LOCATIONS:
Locations (1):
- California Center for Sleep Disorders, Alameda, California, United States

IPD SHARING:
Plan to Share IPD: No